CLINICAL TRIAL: NCT03768453
Title: EARLY-MYO-CMR (EARLY Assessment of MYOcardial Tissue Characteristics by CMR in STEMI) Registry
Brief Title: EARLY-MYO-CMR Registry
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: RenJi Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: EARLY-MYO-CMR
Record Dates: First submitted 2018-12-03; First posted 2018-12-07 (Actual); Last update posted 2020-06-23 (Actual); Status verified 2019-06

CONDITIONS: ST-segment Elevation Myocardial Infarction (STEMI)
MeSH Terms: conditions — ST Elevation Myocardial Infarction

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: None Retained — Routine blood test includes CBC, Liver&Renal function, VBG, cardiac enzymes, glucose, serum lipid etc.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this registry is to depict the myocardial tissue characteristics in STEMI patients by CMR and other cardiac imaging modalities and to assess the prognostic value of imaging-derived indices. Information will be collected prospectively in about 1000 STEMI patients in 10 sites. Subjects will be followed for up to 5 years.

DETAILED DESCRIPTION:
This is a prospective, multi-center, non-randomized, observational registry study of STEMI patients that undergo CMR examination. Information of other cardiac imagings and clinical outcomes are also prospectively collected in the database. This project will establish a prospective registry of 1000 STEMI patients in 10 sites with follow-ups of up to 5 years.

The aim of the project will be as following:

1. To investigate myocardial tissue features and functional changes in STEMI patients.
2. To identify CMR-derived indices that are associated with adverse clinical outcomes.
3. To compare CMR with other alternative cardiac imaging modalities (i.e., echocardiography or SPECT) on prognostic prediction in STEMI patients.
4. To compare myocardial tissue characteristics and functional changes in STEMI and NSTEMI patients (data derived from EARLY-MYO-CMR II Registry).

ELIGIBILITY:
Inclusion Criteria:

STEMI patients who have had CMR imaging performed and have provided written consent.

1. Patents older than 18 years old with myocardial infarction diagnosed by:

   1. typical ischemic symptom,
   2. New ischaemic ECG changes;: ≥2 mm ST-segment elevation in 2 contiguous precordial leads or ≥1 mm ST-segment elevation in 2 contiguous extremity leads ;
   3. elevated cardiac troponin value with at least one value above 99th percentile upper reference limit(UPL);
   4. confirmed by coronary angiography (CAG) or imaging evidence of new loss of viable myocardium or new regional wall motion abnormality in a pattern consistent with an ischaemic aetiology.
2. Patients who have had CMR imaging performed and have agreed to comply with the follow up requirements.

Exclusion Criteria:

1. Patient who is unable to comply with the follow-up schedule.
2. Patient who has any medical conditions that in the opinion of the investigators will not be appropriate to participate in the study.
3. Patient has a life expectancy of less than 6 months due to any condition.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: STEMI patients undergo CMR examination are eligible for this registry.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2012-05-08 (Actual); Primary Completion 2020-07-08 (Estimated); Study Completion 2020-12-01 (Estimated)

PRIMARY OUTCOMES:
Major adverse cardiac events | 1 year
  MACE

CONTACTS AND LOCATIONS:
Overall Officials: Jun Pu, Principal Investigator — Renji Hospital, School of Medicine, Shanghai Jiaotong University.
Locations (1):
- Ren Ji Hospital Affliated to School of Medicine, Shanghai Jiao Tong University, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Derived] Dong JX, Wei L, Jin LX, He J, Zhao CX, Ding S, Kong LC, Yang F, An DA, Wu CW, Chen BH, Wang HW, Yang YN, Ge H, Pu J. MR Uniformity Ratio Estimates to Evaluate Ventricular Mechanical Dyssynchrony and Prognosis After ST-Segment Elevation Myocardial Infarction. J Magn Reson Imaging. 2024 May;59(5):1820-1831. doi: 10.1002/jmri.28998. Epub 2023 Oct 13. PMID 37830268
- [Derived] Lai W, Chen-Xu Z, Jian-Xun D, Jie H, Ling-Cong K, Dong-Ao-Lei A, Bing-Hua C, Song D, Zheng L, Fan Y, Hu-Wen W, Jian-Rong X, Heng G, Jun P. Prognostic implications of left ventricular torsion measured by feature-tracking cardiac magnetic resonance in patients with ST-elevation myocardial infarction. Eur Heart J Cardiovasc Imaging. 2023 May 31;24(6):785-795. doi: 10.1093/ehjci/jeac177. PMID 36056877
- [Derived] Zhao Y, Lu X, Wan F, Gao L, Lin N, He J, Wei L, Dong J, Qin Z, Zhong F, Qiao Z, Wang W, Ge H, Ding S, Yang Y, Xiu J, Shan P, Yan F, Zhao S, Ji Y, Pu J. Disruption of Circadian Rhythms by Shift Work Exacerbates Reperfusion Injury in Myocardial Infarction. J Am Coll Cardiol. 2022 May 31;79(21):2097-2115. doi: 10.1016/j.jacc.2022.03.370. PMID 35618347
- [Derived] Lai W, Jie H, Jian-Xun D, Ling-Cong K, Jun-Tong Z, Bo-Zhong S, Dong-Ao-Lei A, Bing-Hua C, Song D, Zheng L, Fan Y, Yi-Ning Y, Fu-Hua Y, Jian-Cheng X, Hu-Wen W, Jian-Rong X, Heng G, Jun P. Impact of Concomitant Impairments of the Left and Right Ventricular Myocardial Strain on the Prognoses of Patients With ST-Elevation Myocardial Infarction. Front Cardiovasc Med. 2021 May 31;8:659364. doi: 10.3389/fcvm.2021.659364. eCollection 2021. PMID 34136542